CLINICAL TRIAL: NCT06239259
Title: Validity and Reliability of Thai Version of Kamath and Stothard Clinical Questionnaire for Diagnosis of Carpal Tunnel Syndrome
Brief Title: Validity and Reliability of Thai Version Clinical Questionnaire for Diagnosis of Carpal Tunnel Syndrome
Status: Recruiting | Type: Observational
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Panai Laohaprasitiporn, MD, Principle investigator, Siriraj Hospital
Other Study IDs: 456/2566(EC4)
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome; Diagnosis; Content validity
MeSH Terms: conditions — Carpal Tunnel Syndrome; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Carpal tunnel syndrome patients: Carpal tunnel syndrome patients
  Interventions: Other: Questionare As described in Secondary Outcomes

INTERVENTIONS:
Other: Questionare As described in Secondary Outcomes — All patients will recieve Questionare As described in Secondary Outcomes, and will be interviewd by a well-trained reaserch assistanced

SUMMARY:
The Kamath and Stothard clinical questionnaire for diagnosing carpal tunnel syndrome (CTS) is a valid score for diagnosis of CTS. However it haven't been translated in to Thai version and the validity and accuracy of the Thai the Thai version have not been yet verified.

The research team recognizes the importance and potential benefits of adapting this assessment for use within the Thai population.Therefore, we aim to conduct this research to translate the questionnaire from the original English to Thai and to assess its validity and reliability for diagnosing patients with Carpal Tunnel Syndrome.

DETAILED DESCRIPTION:
Carpal Tunnel Syndrome is a common condition among working and older adults. The incidence of the disease ranges from 7 to 19 percent in the general population, with an approximate rate of 99 cases per 100,000 population per year. Symptoms are typically associated with hand and wrist function. Patients frequently seek medical attention due to numbness or pain in their hands after prolonged, continuous use. Some individuals may experience persistent numbness or pain in their hands, significantly impacting their daily lives. In cases of prolonged symptoms, weakness of the thumb may also occur.

The diagnosis is established through a comprehensive history and physical examination, with symptoms including numbness in the thumb and index finger, as well as the middle finger and the portion of the ring finger adjacent to the middle finger. Some individuals may experience pain, especially at night or in cold conditions, often aggravated by the use of the hands and wrists. The physical examination reveals a reduction in tactile sensations in the regions corresponding to the thumb, index finger, middle finger, and half of the ring finger near the middle finger. In severe cases, weakness of the abductor pollicis brevis muscle or muscle atrophy in the thenar area may be detected. Confirmation of the diagnosis can be achieved through an electrodiagnostic study of muscles and nerves.

Kamath and Stothard clinical questionnaire was developed to help clinician in the diagnosis of CTS, with score more than 5 the diagnosis can be achieve without needed for further electrodiagnostic test. However it haven't been translated in to Thai version and the validity and accuracy of the Thai the Thai version have not been yet verified.

The research team recognizes the importance and potential benefits of adapting this assessment for use within the Thai population.Therefore, we aim to conduct this research to translate the questionnaire from the original English to Thai and to assess its validity and reliability for diagnosing patients with Carpal Tunnel Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older who are admitted to Siriraj Hospital with signs and symptoms consistent with carpal tunnel disease.
* Diagnosis of carpal tunnel disease was confirm with electrodiagnostic study and electromyography
* Must be able to communicate in Thai.

Exclusion Criteria:

* Patients diagnosed with other neurological diseases such as cerebrovascular disease, cervical radiculopathy, diabetic neuropathy, tumors of the nerve endings in the arm, and other peripheral neuropathy.
* Pregnancy or breastfeeding
* History of recieving chemotheraphy agent
* Patient who recieved surgical treatment for carpal tunnel syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Carpal tunnel syndrome patients who recieved conservative treatment at Single-center, Siriraj hospital, Thailand
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Validity of Thai version of Kamath and Stothard Questionnaire in carpal tunnel syndrome patients | Pre-treatment
  The questionnaire composes of 9 clinical questions asking whether the patient has any symptom of carpal tunnel syndrome. The total score is the sum of the score from each question. Total score ranges from -2 to 11. Higher scores indicate a greater probability of the condition, prompting further investigation and potential referral to a specialist.
  Concurrent validity is evaluated by comparing this questionnaire with the Boston carpal tunnel questionnaire.
Reliability of Thai version of Kamath and Stothard Questionnaire in carpal tunnel syndrome patients | Pre-treatment and 2 weeks later
  The questionnaire composes of 9 clinical questions asking whether the patient has any symptom of carpal tunnel syndrome. The total score is the sum of the score from each question. Total score ranges from -2 to 11. Higher scores indicate a greater probability of the condition, prompting further investigation and potential referral to a specialist.
  Intra-observer reliability is measured using Kappa statistics for each answered question between two different periods.

SECONDARY OUTCOMES:
Thai version of Boston carpal tunnel questionnaire (BCTQ) | Pre-treatment
  This questionnaire designed to assess the severity of carpal tunnel syndrome. It consists of two parts:
  Part 1 involves the evaluation of hand abnormalities, comprising 11 items (symptom severity score).
  Part 2 assesses the loss of hand function and includes another 8 items (function severity score).
  Symptom Severity Scale (SSS): The scores for each item are averaged to provide a mean score, ranging from 1-5. Higher scores indicate more severe symptoms.
  Functional Status Scale (FSS): The scores for each item are averaged to provide a mean score, ranging from 1-5. Higher scores indicate greater difficulty in performing daily activities.
Thai version of EQ-5D-5L questionaire | Pre-treatment
  This questionnaire comprises of two parts:
  Part 1, consisting of 5 questions about supervision, self-care, normal activities, medical/discomfort, and coldness/depression. The questions related to medical/discomfort and coldness/depression have 5 options each.
  Part 2, directly assessing health conditions on a visual analog scale from 0 to 100. Here, 0 represents the most adverse change in health, and 100 represents the most positive change in health.
Thai version of Patient-rated wrist evaluation questionaire (PRWE) | Pre-treatment
  This tool use to assess the functional ability of the wrist. The tool consists of two parts: pain and the ability to perform activities.
  Part 1: Pain subscale comprises a total of 5 questions, each with multiple-choice answers ranging from 0 to 10 points. A score of 0 indicates no pain, while 10 points indicate the most intense or constant pain.
  Part 2: Function subscale includes a total of 10 questions related to daily activities, characterized on a scale from 0 to 10. A score of 0 indicates no interference with daily activities, while 10 points indicate significant interference and limitations in daily living.
  The pain subscale has a maximum total score of 50 and the function subscale has a maximum total score of 100. A higher score reflects more pain or greater difficulty in performing the activities. The total score for the PRWE is obtained from a summation of the total pain subscale and half of the total function subscale.
Thai version of Quick Disabilities of Arm, Shoulder and Hand questionaire (QuickDASH) | Pre-treatment
  The QuickDASH (Quick Disabilities of the Arm, Shoulder, and Hand) is a shortened version of the original DASH questionnaire, designed to measure physical function and symptoms in people with musculoskeletal disorders of the upper limb. It consists of 11 items. Patients rate their difficulty or severity of symptoms over the past week on a scale from 1 (no difficulty) to 5 (unable to perform).
  The average score is the sum of responded items divided by number of completed items. Then, the average score is transform to a 0-100 scale by subtracting the average score with 1 and divided by 4 and then multiply with 25.
Thai Language of the Neuropathic Pain Diagnostic Questionnaire (DN4) | Pre-treatment
  This is a 10-item questionnaire designed to detect neuropathic pain has been translated and validated in the Thai version. It consists of 2 parts:
  Part 1 is a section with patient interview questions comprising 7 yes or no questions. Each 'yes' answer is scored as 1 point and 'no' answer is scored as 0 point.
  Part 2 is the physical examination section with 3 questions, and each affirmative finding is scored as 1 point.
  The test has a total score of 10 points, ranging from 0 to 10. The highest score possible is 10 points, while the lowest score is 0 points.
  A total score of >4 points indicates pain resulting from a neurological disorder, specifically neuropathic pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferry S, Pritchard T, Keenan J, Croft P, Silman AJ. Estimating the prevalence of delayed median nerve conduction in the general population. Br J Rheumatol. 1998 Jun;37(6):630-5. doi: 10.1093/rheumatology/37.6.630. PMID 9667616
- [Background] von Schroeder HP, Botte MJ. Carpal tunnel syndrome. Hand Clin. 1996 Nov;12(4):643-55. PMID 8953285
- [Background] Newington L, Harris EC, Walker-Bone K. Carpal tunnel syndrome and work. Best Pract Res Clin Rheumatol. 2015 Jun;29(3):440-53. doi: 10.1016/j.berh.2015.04.026. Epub 2015 May 27. PMID 26612240
- [Background] Levine DW, Simmons BP, Koris MJ, Daltroy LH, Hohl GG, Fossel AH, Katz JN. A self-administered questionnaire for the assessment of severity of symptoms and functional status in carpal tunnel syndrome. J Bone Joint Surg Am. 1993 Nov;75(11):1585-92. doi: 10.2106/00004623-199311000-00002. PMID 8245050
- [Background] Upatham S, Kumnerddee W. Reliability of Thai version Boston questionnaire. J Med Assoc Thai. 2008 Aug;91(8):1250-6. PMID 18788699
- [Background] Kamath V, Stothard J. A clinical questionnaire for the diagnosis of carpal tunnel syndrome. J Hand Surg Br. 2003 Oct;28(5):455-9. doi: 10.1016/s0266-7681(03)00151-7. PMID 12954256
- [Background] Bonett DG. Sample size requirements for estimating intraclass correlations with desired precision. Stat Med. 2002 May 15;21(9):1331-5. doi: 10.1002/sim.1108. PMID 12111881
- [Background] Kimman M, Vathesatogkit P, Woodward M, Tai ES, Thumboo J, Yamwong S, Ratanachaiwong W, Wee HL, Sritara P. Validity of the Thai EQ-5D in an occupational population in Thailand. Qual Life Res. 2013 Aug;22(6):1499-506. doi: 10.1007/s11136-012-0251-2. Epub 2012 Aug 25. PMID 22926727
- [Background] Laohaprasitiporn P, Monteerarat Y, Jaderojananont W, Limthongthang R, Vathana T. Validity, Reliability and Responsiveness of the Thai Version of Patient-Rated Wrist Evaluation (Th-PRWE) in Distal Radius Fracture Patients. Siriraj Medical Journal. 2021;73(4):275-81.
- [Background] Bonett, DG, Wright, TA. Cronbach's alpha reliability: Interval estimation, hypothesis testing, and sample size planning. J Organiz Behav 2015; 36: 3-15.
- [Background] Shoukri MM, Asyali MH, Donner A. Design of reliability study. Statistical Methods in Medical Research 2004; 13: 251-71.
- [Background] Tongprasert S, Rapipong J, Buntragulpoontawee M. The cross-cultural adaptation of the DASH questionnaire in Thai (DASH-TH). J Hand Ther. 2014 Jan-Mar;27(1):49-54. doi: 10.1016/j.jht.2013.08.020. Epub 2013 Oct 5. PMID 24100056
- [Background] Chaudakshetrin P, Prateepavanich P, Chira-Adisai W, Tassanawipas W, Leechavengvongs S, Kitisomprayoonkul W. Cross-cultural adaptation to the Thai language of the neuropathic pain diagnostic questionnaire (DN4). J Med Assoc Thai. 2007 Sep;90(9):1860-5. PMID 17957931